CLINICAL TRIAL: NCT06707701
Title: Correlation Among Various OLGA and OLGIM Stages, Digestive Symptom Scores, and Acupuncture Treatment in Patients with Chronic Atrophic Gastritis:a Multicenter Cross-sectional Pilot Survey
Brief Title: Correlation Among Various OLGA and OLGIM Stages, Digestive Symptom Scores, and Acupuncture Treatment in Patients with Chronic Atrophic Gastritis
Status: Not yet recruiting | Type: Observational
Sponsor: Yi Liang (Other)
Collaborators: Zhejiang Provincial Department of Science and Technology (Unknown)
Responsible Party: Sponsor-Investigator, Yi Liang, Research Fellow, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Other Study IDs: 20241102100617911
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Chronic Atrophic Gastritis (CAG)
Keywords: chronic atrophic gastritis; global overall symptom scale; serum pepsinogen; operative link for gastritis assessment; operative link for gastric intestinal metaplasia assessment
MeSH Terms: conditions — Gastritis, Atrophic | interventions — Acupuncture Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum pepsinogen extracted and detected in venous blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: acupuncture — Whether or not a patient has been treated with acupuncture will be one of the exposure factors of interest in the study

SUMMARY:
Brief Summary Template for the Study:

The goal of this observational study is to examine the relationship between digestive symptom scores, serum pepsinogen indices, and histopathological OLGA and OLGIM systematic staging of the gastric mucosa in patients with chronic atrophic gastritis(CAG), aiming to determine the degree of correlation between clinical manifestations, non-invasive laboratory tests, and the gold standard of diagnostic histopathology.To evaluate the comprehensive therapy, readiness and acceptance of acupuncture, utilization rates of various acupuncture therapies, self-assessed efficacy of acupuncture, and endoscopic histopathological alterations in patients with CAG.According to the aforementioned study, it is anticipated to enhance the optimization of acupuncture clinical research protocols for chronic atrophic gastritis, improve treatment efficacy, and offer more effective and rational therapy alternatives for patients.The main question it aims to answer is:

To determine if the outcomes of combined serologic testing of symptoms in patients with CAG can serve as a method for monitoring disease development and if long-term follow-up can be supported？

A group of participants with recorded GI symptom scores and blood pepsinogen levels will respond to online survey questions regarding the severity of their chronic atrophic gastritis progression over the course of 1 year.

DETAILED DESCRIPTION:
This study is a multicenter cross-sectional pilot survey

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the diagnostic criteria for chronic atrophic gastritis;
* Individuals aged 18 to 75 years, irrespective of gender;
* Capable of comprehending and consenting to participate in this study by signing the informed consent form.

Exclusion Criteria:

* Autoimmune gastritis (type A chronic atrophic gastritis);
* Patients diagnosed with Gastroesophageal Reflux Disease (GERD) by endoscopy or other examinations or patients diagnosed with high-grade intraepithelial neoplasia by upper gastrointestinal endoscopy and gastric mucosal biopsy pathology;
* Patients with confirmed or unable to exclude malignant tumors, especially esophageal and gastric cancers; patients with other upper gastrointestinal tract pathologies such as peptic ulcer or Barrett's esophagus;
* Those who cannot complete the questionnaire due to unconsciousness, inability to communicate normally or other reasons; those with incomplete information.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involved the recruitment of CAG patients from endoscopy centers, outpatient clinics, and inpatient clinics within the Department of Splenology and Gastroenterology at Zhongshan Hospital in Zhejiang Province, designated as the primary recruitment center, along with the First People's Hospital of Hangzhou and Hangzhou Hospital of Traditional Chinese Medicine as secondary recruitment centers.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between gastrointestinal symptom scores combined with serum pepsinogen indexes and histopathologic OLGA and OLGIM systematic staging of gastric mucosa in patients with CAG | Gastroscopy and pathology reports within one year, serology and symptom assessment within one week of participant enrollment
  The investigators gathered clinical data on the overall condition, occupation, personal history, family history, H. pylori infection, gastrointestinal symptom scores, serum pepsinogen index, gastroscopy reports, pathological findings, and other biological characteristics of CAG patients, along with data pertaining to acupuncture treatment. The investigators then analyzed the correlation between the gastrointestinal symptom scores, the serum pepsinogen index, and the gastric mucosal histopathology OLGA and OLGIM. The investigators examined the relationship between gastrointestinal symptom scores, serum pepsinogen levels, and the histopathological OLGA and OLGIM stages of gastric mucosa to determine the correlation between clinical manifestations, non-invasive laboratory tests, and the definitive diagnostic standard of histopathology, thereby offering support for clinicians.

SECONDARY OUTCOMES:
Correlation coefficients of relevant exposure factors (including acupuncture treatment status) with OLGA, OLGIM pathologic stage and GI symptom score, respectively | Patient's treatment to date after diagnosis of chronic atrophic gastritis, and whether participant has received acupuncture in the last 3 months
  With the goal of further optimizing the clinical research protocols of acupuncture for CAG, improving the therapeutic effects, and offering a more effective and affordable treatment option for patients with chronic atrophic gastritis, the investigators examined the overall treatment of CAG patients, willingness and acceptance of acupuncture treatment, application rate of various acupuncture therapies, self-perceived acupuncture efficacy, and endoscopic histopathological changes.

CONTACTS AND LOCATIONS:
Locations (1):
- the Ethics Board of The Third Affiliated Hospital of Zhejiang Chinese Medicinal University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF